CLINICAL TRIAL: NCT03340519
Title: Early MRI Prediction of Response to Medical Therapy and Mucosal Healing in Small Bowel Crohn's Disease
Brief Title: Early MRI Prediction of Crohns
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN_EarlyMRCrohns
Record Dates: First submitted 2017-11-09; First posted 2017-11-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease
Keywords: Crohn; MRI
MeSH Terms: conditions — Crohn Disease | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Healthy Controls: Healthy Controls will undergo MR imaging to optimize MR techniques for bowel assessment and to acquire normative data
  Interventions: Device: MR Imaging
- Newly Diagnosed Crohns Patients: MR imaging will be performed in newly diagnosed CD patients prior to initiation of infliximab therapy in order to obtain baseline measures in the setting of active intestinal inflammation
  Interventions: Device: MR Imaging

INTERVENTIONS:
Device: MR Imaging — Novel MR imaging will be performed to provide bowel anatomic and functional data

SUMMARY:
The investigators plan a prospective study designed to optimize and translate noncontrast, novel Magnetic Resonance Imaging (MRI) techniques for detecting and measuring intestinal inflammation as well as for allowing early prediction of response to medical therapy in small bowel Crohn's Disease (CD).

DETAILED DESCRIPTION:
The investigators plan to evaluate novel MRI techniques to measure: 1) mesenteric/intestinal blood flow using phase-contrast cine MRI, 2) intestinal motility (peristalsis) using dynamic cine MRI, and 3) bowel wall perfusion and molecular water diffusion. Precise objective measurements of diseased bowel blood flow (in ml/min) and bowel motility (in contractions per minute) are not currently used in the clinical care of CD patients, while diffusion-weighted imaging is typically used in a qualitative manner. None of these techniques have been evaluated for predicting eventual response to therapy or correlated with endoscopic mucosal healing in pediatric or adult CD.

ELIGIBILITY:
Inclusion Criteria:

Healthy Control Group

-Be able to tolerate up to 45 minutes in an MRI scanner

Newly Diagnosed Crohns Group

* Newly diagnosed, pathology-confirmed diagnosis of small bowel Crohn's disease,
* Expected to receive infliximab (Remicade; Janssen Biotech, Inc.) or other anti-Tumor Necrosis Factor (anti-TNF) medical therapy,
* Between 11 to 25 years of age and able to assent/consent,
* Be available for follow-up MRI at 4-weeks and 6-months after the initiation of treatment,
* Be able to tolerate up to 45 minutes in an MRI scanner.

Exclusion Criteria:

Healthy Control Group

* Inability to obtain assent/consent,
* Inability to tolerate 45 minutes in an MRI scanner,
* Contraindication to MRI (e.g., MRI incompatible implant or support device),
* Previous (remote) diagnosis or treatment of inflammatory bowel disease or other intestinal disease,
* History of intra-abdominal surgery, including surgery on the intestine,
* Pregnancy. Point-of-care urine pregnancy testing will be performed on all female study participants of reproductive potential (pediatric and adult) prior to each research MRI exam.

Newly Diagnosed Crohns Group

* Inability to obtain assent/consent,
* Inability to tolerate 45 minutes in an MRI scanner,
* Contraindication to MRI (e.g., MRI incompatible implant or support device),
* Previous (remote) diagnosis or treatment of inflammatory bowel disease,
* History of intra-abdominal surgery, including surgery on the intestine,
* Known bleeding disorder/coagulopathy (contraindication for adult subjects, as this may increase the risk of research colonoscopy),
* Pregnancy. Point-of-care urine pregnancy testing will be performed on all female study participants of reproductive potential (pediatric and adult) prior to each research MRI exam.

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy Control Group General population Newly Diagnosed Crohns Group Cincinnati Children's Inflammatory Bowel Disease Clinic
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
Prediction of therapeutic response in patients with Crohns disease | 30 minutes
  Assess novel MRI techniques for ability to predict early response to infliximab therapy in 20 newly diagnosed small bowel CD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan R Dillman, MD, MSc, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified data will be shared

REFERENCES:
- [Background] Peyrin-Biroulet L, Loftus EV Jr, Colombel JF, Sandborn WJ. The natural history of adult Crohn's disease in population-based cohorts. Am J Gastroenterol. 2010 Feb;105(2):289-97. doi: 10.1038/ajg.2009.579. Epub 2009 Oct 27. PMID 19861953
- [Background] Aggarwal D, Limdi JK. Anti-TNF therapy is associated with a reduction in radiation exposure in patients with Crohn's disease. Eur J Gastroenterol Hepatol. 2015 Jan;27(1):13-9. doi: 10.1097/MEG.0000000000000222. PMID 25341058
- [Background] Church PC, Guan J, Walters TD, Frost K, Assa A, Muise AM, Griffiths AM. Infliximab maintains durable response and facilitates catch-up growth in luminal pediatric Crohn's disease. Inflamm Bowel Dis. 2014 Jul;20(7):1177-86. doi: 10.1097/MIB.0000000000000083. PMID 24865777
- [Background] Hyams JS, Lerer T, Griffiths A, Pfefferkorn M, Kugathasan S, Evans J, Otley A, Carvalho R, Mack D, Bousvaros A, Rosh J, Mamula P, Kay M, Crandall W, Oliva-Hemker M, Keljo D, LeLeiko N, Markowitz J; Pediatric Inflammatory Bowel Disease Collaborative Research Group. Long-term outcome of maintenance infliximab therapy in children with Crohn's disease. Inflamm Bowel Dis. 2009 Jun;15(6):816-22. doi: 10.1002/ibd.20845. PMID 19107783
- [Background] Kane SV, Jaganathan S, Bedenbaugh AV, Palmer L, Schwartz DA. Anti-tumor necrosis factor agents reduce corticosteroid use compared with azathioprine in patients with Crohn's disease. Curr Med Res Opin. 2014 Sep;30(9):1821-6. doi: 10.1185/03007995.2014.928273. Epub 2014 Jun 2. PMID 24884302
- [Background] Mandel MD, Miheller P, Mullner K, Golovics PA, Lakatos PL. Have biologics changed the natural history of Crohn's disease? Dig Dis. 2014;32(4):351-9. doi: 10.1159/000358135. Epub 2014 Jun 23. PMID 24969279
- [Background] Viola F, Civitelli F, Di Nardo G, Barbato MB, Borrelli O, Oliva S, Conte F, Cucchiara S. Efficacy of adalimumab in moderate-to-severe pediatric Crohn's disease. Am J Gastroenterol. 2009 Oct;104(10):2566-71. doi: 10.1038/ajg.2009.372. Epub 2009 Jun 23. PMID 19550415
- [Background] Walters TD, Kim MO, Denson LA, Griffiths AM, Dubinsky M, Markowitz J, Baldassano R, Crandall W, Rosh J, Pfefferkorn M, Otley A, Heyman MB, LeLeiko N, Baker S, Guthery SL, Evans J, Ziring D, Kellermayer R, Stephens M, Mack D, Oliva-Hemker M, Patel AS, Kirschner B, Moulton D, Cohen S, Kim S, Liu C, Essers J, Kugathasan S, Hyams JS; PRO-KIIDS Research Group. Increased effectiveness of early therapy with anti-tumor necrosis factor-alpha vs an immunomodulator in children with Crohn's disease. Gastroenterology. 2014 Feb;146(2):383-91. doi: 10.1053/j.gastro.2013.10.027. Epub 2013 Oct 23. PMID 24162032
- [Background] Dillman JR, Adler J, Zimmermann EM, Strouse PJ. CT enterography of pediatric Crohn disease. Pediatr Radiol. 2010 Jan;40(1):97-105. doi: 10.1007/s00247-009-1465-5. Epub 2009 Nov 20. PMID 19936733
- [Background] Mollard BJ, Smith EA, Dillman JR. Pediatric MR enterography: technique and approach to interpretation-how we do it. Radiology. 2015 Jan;274(1):29-43. doi: 10.1148/radiol.14122449. PMID 25531478
- [Background] Brenner DJ. Should computed tomography be the modality of choice for imaging Crohn's disease in children? The radiation risk perspective. Gut. 2008 Nov;57(11):1489-90. doi: 10.1136/gut.2008.156265. No abstract available. PMID 18941001
- [Background] Brenner DJ, Hall EJ. Computed tomography--an increasing source of radiation exposure. N Engl J Med. 2007 Nov 29;357(22):2277-84. doi: 10.1056/NEJMra072149. No abstract available. PMID 18046031
- [Background] McDonald RJ, McDonald JS, Kallmes DF, Jentoft ME, Murray DL, Thielen KR, Williamson EE, Eckel LJ. Intracranial Gadolinium Deposition after Contrast-enhanced MR Imaging. Radiology. 2015 Jun;275(3):772-82. doi: 10.1148/radiol.15150025. Epub 2015 Mar 5. PMID 25742194
- [Background] Ramalho J, Castillo M, AlObaidy M, Nunes RH, Ramalho M, Dale BM, Semelka RC. High Signal Intensity in Globus Pallidus and Dentate Nucleus on Unenhanced T1-weighted MR Images: Evaluation of Two Linear Gadolinium-based Contrast Agents. Radiology. 2015 Sep;276(3):836-44. doi: 10.1148/radiol.2015150872. Epub 2015 Jun 16. PMID 26079490
- [Background] Bouguen G, Levesque BG, Feagan BG, Kavanaugh A, Peyrin-Biroulet L, Colombel JF, Hanauer SB, Sandborn WJ. Treat to target: a proposed new paradigm for the management of Crohn's disease. Clin Gastroenterol Hepatol. 2015 Jun;13(6):1042-50.e2. doi: 10.1016/j.cgh.2013.09.006. Epub 2013 Sep 10. PMID 24036054
- [Background] Shah SC, Colombel JF, Sands BE, Narula N. Systematic review with meta-analysis: mucosal healing is associated with improved long-term outcomes in Crohn's disease. Aliment Pharmacol Ther. 2016 Feb;43(3):317-33. doi: 10.1111/apt.13475. Epub 2015 Nov 25. PMID 26607562
- [Background] Reinink AR, Lee TC, Higgins PD. Endoscopic Mucosal Healing Predicts Favorable Clinical Outcomes in Inflammatory Bowel Disease: A Meta-analysis. Inflamm Bowel Dis. 2016 Aug;22(8):1859-69. doi: 10.1097/MIB.0000000000000816. PMID 27206015
- [Background] Nayak KS, Nielsen JF, Bernstein MA, Markl M, D Gatehouse P, M Botnar R, Saloner D, Lorenz C, Wen H, S Hu B, Epstein FH, N Oshinski J, Raman SV. Cardiovascular magnetic resonance phase contrast imaging. J Cardiovasc Magn Reson. 2015 Aug 9;17(1):71. doi: 10.1186/s12968-015-0172-7. PMID 26254979
- [Background] Heiss SG, Li KC. Magnetic resonance angiography of mesenteric arteries. A review. Invest Radiol. 1998 Sep;33(9):670-81. doi: 10.1097/00004424-199809000-00023. PMID 9766052
- [Background] Akerman A, Mansson S, Fork FT, Leander P, Ekberg O, Taylor S, Menys A, Ohlsson B. Computational postprocessing quantification of small bowel motility using magnetic resonance images in clinical practice: An initial experience. J Magn Reson Imaging. 2016 Aug;44(2):277-87. doi: 10.1002/jmri.25166. Epub 2016 Jan 23. PMID 26801196
- [Background] Bickelhaupt S, Pazahr S, Chuck N, Blume I, Froehlich JM, Cattin R, Raible S, Bouquet H, Bill U, Rogler G, Frei P, Boss A, Patak MA. Crohn's disease: small bowel motility impairment correlates with inflammatory-related markers C-reactive protein and calprotectin. Neurogastroenterol Motil. 2013 Jun;25(6):467-73. doi: 10.1111/nmo.12088. Epub 2013 Mar 18. PMID 23495824
- [Background] Froehlich JM, Waldherr C, Stoupis C, Erturk SM, Patak MA. MR motility imaging in Crohn's disease improves lesion detection compared with standard MR imaging. Eur Radiol. 2010 Aug;20(8):1945-51. doi: 10.1007/s00330-010-1759-x. Epub 2010 Apr 9. PMID 20379822
- [Background] Menys A, Atkinson D, Odille F, Ahmed A, Novelli M, Rodriguez-Justo M, Proctor I, Punwani S, Halligan S, Taylor SA. Quantified terminal ileal motility during MR enterography as a potential biomarker of Crohn's disease activity: a preliminary study. Eur Radiol. 2012 Nov;22(11):2494-501. doi: 10.1007/s00330-012-2514-2. Epub 2012 Jun 3. PMID 22661057
- [Background] Chenevert TL, Sundgren PC, Ross BD. Diffusion imaging: insight to cell status and cytoarchitecture. Neuroimaging Clin N Am. 2006 Nov;16(4):619-32, viii-ix. doi: 10.1016/j.nic.2006.06.005. PMID 17148023
- [Background] Ream JM, Dillman JR, Adler J, Khalatbari S, McHugh JB, Strouse PJ, Dhanani M, Shpeen B, Al-Hawary MM. MRI diffusion-weighted imaging (DWI) in pediatric small bowel Crohn disease: correlation with MRI findings of active bowel wall inflammation. Pediatr Radiol. 2013 Sep;43(9):1077-85. doi: 10.1007/s00247-013-2712-3. Epub 2013 Aug 16. PMID 23949929
- [Background] Dillman JR, Smith EA, Sanchez R, Adler J, Fazeli S, Zhang B, Davenport MS. DWI in Pediatric Small-Bowel Crohn Disease: Are Apparent Diffusion Coefficients Surrogates for Disease Activity in Patients Receiving Infliximab Therapy? AJR Am J Roentgenol. 2016 Nov;207(5):1002-1008. doi: 10.2214/AJR.16.16477. Epub 2016 Aug 9. PMID 27505635
- [Background] Le Bihan D, Breton E, Lallemand D, Grenier P, Cabanis E, Laval-Jeantet M. MR imaging of intravoxel incoherent motions: application to diffusion and perfusion in neurologic disorders. Radiology. 1986 Nov;161(2):401-7. doi: 10.1148/radiology.161.2.3763909.
- [Background] Freiman M, Perez-Rossello JM, Callahan MJ, Bittman M, Mulkern RV, Bousvaros A, Warfield SK. Characterization of fast and slow diffusion from diffusion-weighted MRI of pediatric Crohn's disease. J Magn Reson Imaging. 2013 Jan;37(1):156-63. doi: 10.1002/jmri.23781. Epub 2012 Aug 24. PMID 22927342
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Hyams JS, Ferry GD, Mandel FS, Gryboski JD, Kibort PM, Kirschner BS, Griffiths AM, Katz AJ, Grand RJ, Boyle JT, et al. Development and validation of a pediatric Crohn's disease activity index. J Pediatr Gastroenterol Nutr. 1991 May;12(4):439-47. PMID 1678008
- [Background] Someya N, Endo MY, Fukuba Y, Hayashi N. Blood flow responses in celiac and superior mesenteric arteries in the initial phase of digestion. Am J Physiol Regul Integr Comp Physiol. 2008 Jun;294(6):R1790-6. doi: 10.1152/ajpregu.00553.2007. Epub 2008 Apr 2. PMID 18385466
- [Background] Mary JY, Modigliani R. Development and validation of an endoscopic index of the severity for Crohn's disease: a prospective multicentre study. Groupe d'Etudes Therapeutiques des Affections Inflammatoires du Tube Digestif (GETAID). Gut. 1989 Jul;30(7):983-9. doi: 10.1136/gut.30.7.983. PMID 2668130
- [Background] Peyrin-Biroulet L, Reinisch W, Colombel JF, Mantzaris GJ, Kornbluth A, Diamond R, Rutgeerts P, Tang LK, Cornillie FJ, Sandborn WJ. Clinical disease activity, C-reactive protein normalisation and mucosal healing in Crohn's disease in the SONIC trial. Gut. 2014 Jan;63(1):88-95. doi: 10.1136/gutjnl-2013-304984. Epub 2013 Aug 23. PMID 23974954